CLINICAL TRIAL: NCT06335316
Title: Effect of Stellate Ganglion Block in Dysphagic Patients With Bulbar Palsy After Ischemic Stroke
Brief Title: Effect of Stellate Nerve Block in Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: wallenburg sym
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Injections; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Nerve Block+ routine rehabilitation treatment (Experimental): The patients were given Nerve block and routine rehabilitation treatment for 10 days.
  Interventions: Procedure: Injection; Drug: Lidocaine Hydrochloride; Behavioral: Comprehensive therapy
- placebo+routine rehabilitation treatment (Placebo Comparator): The patients were given placebo block and routine rehabilitation treatment for 10 days.
  Interventions: Behavioral: Comprehensive therapy; Behavioral: placebo

INTERVENTIONS:
Procedure: Injection — The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Stellate Nerve Block+ routine rehabilitation treatment
Drug: Lidocaine Hydrochloride — the patients were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g)
  Arms: Stellate Nerve Block+ routine rehabilitation treatment
Behavioral: Comprehensive therapy — All the participants are provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.).
Behavioral: placebo — The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck. Only normal saline was used
  Arms: placebo+routine rehabilitation treatment

SUMMARY:
This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in China. Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment,Yale Pharyngeal Residue Severity Rating Scale, video fluoroscopic swallowing study (VFSS), Functional Oral Intake Scale, and penetration-aspiration scale (PAS) were used to assess swallowing function.

DETAILED DESCRIPTION:
Dysphagia is a frequent and potentially serious complication of stroke. This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in China. Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment,Yale Pharyngeal Residue Severity Rating Scale, video fluoroscopic swallowing study (VFSS), Functional Oral Intake Scale, and penetration-aspiration scale (PAS) were used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke according to the diagnostic criteria, with the stroke occurring in the medulla oblongata and diagnosed as bulbar palsy.
* Dysphagia.
* Age >18 years.
* First-time stroke.
* Steady vital signs,
* Transferred or admitted to the Department of Rehabilitation Medicine within 15d after onset.

Exclusion Criteria:

* Allergy to Lidocaine injection or vitamin B12 injection;
* Severe cognitive impairment;
* Coagulation disorders;
* Severe dysfunction of organs including heart, lungs, kidney, liver, etc.;
* Complicated with other neurological diseases;
* Dysphagia caused by other diseases or reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 10
  The Functional Oral Intake Scale (FOIS) is a tool used to assess the level of independence in oral intake for individuals with swallowing difficulties. The scale ranges from Level 1 to Level 7, with higher Levels indicating better swallowing function.

SECONDARY OUTCOMES:
Yale Pharyngeal Residue Severity Rating Scale | day 1 and day 10
  The Yale Pharyngeal Residue Severity Rating Scale (Yale) was used to assess the severity of pharyngeal residue in patients. While PAS primarily evaluated whether food or liquid entered the airway, Yale focused on the condition of pharyngeal residue. The scale includes the four levels from 0 to 3, with lower levels indicating less severe pharyngeal residue.
penetration-aspiration scale | day 1 and day 10
  this assessment evaluated the patient's swallowing of contrast medium and whether there was retention, penetration, and aspiration. It included multiple items, each with the corresponding criteria, Specifically, whether the swallowed material entered the airway, passed through or contacted the vocal cords, and whether the patient exhibited the corresponding ability to clear. There were 8 levels in the results, with higher levels indicating more severe aspiration.
The Swallowing Quality of Life Questionnaire | day 1 and day 10
  The Swallowing Quality of Life Questionnaire (SWAL-QOL) is a tool designed to assess how swallowing difficulties impact an individual's quality of life. The questionnaire covers various aspects such as eating, speech, and social interaction to understand the challenges and effects of swallowing disorders on daily life.
  SWAL-QOL scores can range from 0 to 100, with higher scores indicating a better quality of life related to swallowing function. Therefore, a higher SWAL-QOL score reflects less negative impact of swallowing difficulties on an individual's overall quality of life, highlighting better adaptation to and management of swallowing issues.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group
Locations (1):
- Huimin Hos., Pengfu, Taiwan